CLINICAL TRIAL: NCT00430105
Title: Randomized Trial of Intravenous Pulse Versus Oral Continuous Cyclophosphamide for Induction of Remission in Systemic ANCA-Associated Vasculitides
Brief Title: Pulse Versus Continuous Cyclophosphamide for Induction of Remission in ANCA-Associated Vasculitides
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC20-CT97-0019; BMH4-CT97-2328; IC20-CT97-0019
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: ANCA Associated Systemic Vasculitis; Wegener's Granulomatosis; Microscopic Polyangiitis
Keywords: Vasculitis; ANCA; Wegener's granulomatosis; Renal vasculitis; Cyclophosphamide
MeSH Terms: conditions — Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Vasculitis | interventions — Cyclophosphamide

INTERVENTIONS:
Drug: cyclophosphamide

SUMMARY:
A comparison of intermittent pulsed cyclophosphamide to daily oral cyclophosphamide for the treatment of ANCA-associated systemic vasculitides with kidney involvement.

Performed by the European Vasculitis Study group.

DETAILED DESCRIPTION:
The primary, ANCA-associated systemic vasculitides (AASV), including Wegener's granulomatosis and microscopic polyangiitis, are progressive, multisystem, autoimmune diseases which respond to immunosuppressive therapy. Their treatment with corticosteroids and cytotoxic drugs has been standardised in a first wave of studies (ECSYSVASTRIAL project), but limitations of such regimens include only partial efficacy and appreciable treatment-related toxicity.

The present trial, CYCLOPS, aims to reduce the cumulative exposure to immunosuppressive drugs by administering cyclophosphamide (CYC) as intermittent pulses. The potential benefit of using CYC in this way for AASV has been demonstrated in preliminary, smaller studies. Patients with previously untreated AASV and, "generalised", but not life threatening, disease with renal involvement, will be randomised to either continuous oral CYC or intermittent pulse CYC. CYC will be continued until three months after remission has been achieved, with a minimum CYC total duration of six months and maximum duration of twelve months; both limbs will then receive the same maintenance regimen of azathioprine and prednisolone.

The study will last 18 months. The primary end-point is the disease-free period, taken as the period of time from remission until relapse or study end; secondary end-points are adverse effects, cumulative damage and immunosuppressive drug exposure. 160 patients will be required.

ELIGIBILITY:
Inclusion Criteria:

1. A new diagnosis of WG, MP or renal-limited vasculitis (RLV) (appendix 5). Patients not previously treated with cytotoxic drugs will be permitted.
2. Renal involvement attributable to active WG, MP or RLV with at least one of the following:

   * elevated serum creatinine between 150 and 500 umol/l.
   * biopsy demonstrating necrotizing glomerulonephritis.
   * red cell casts.
   * haematuria with >30 red blood cells/high powered field and proteinuria > 1g/24hr.
3. ANCA positivity or confirmatory histology or both (appendix 5). ANCA positivity requires a typical CANCA pattern by indirect immunofluorescence (IIF), (preferably confirmed by anti-PR3 ELISA), or the presence of PR3-ANCA or MPO-ANCA determined by ELISA, PANCA requires confirmation by anti-MPO ELISA [6]. (Central review of ANCA serology and histology will be performed).
4. Age 18-80 years.

Exclusion Criteria:

1. More than two weeks treatment with cyclophosphamide (CYC) or other cytotoxic drug within previous year or with oral corticosteroids (OCS) for more than 4 weeks. If the patient has received >1.0g of methyl-prednisolone prior to the study start, discuss with trial co-ordinator.
2. Co-existence of another multisystem autoimmune disease, e.g. SLE.
3. Hepatitis Be antigen positive or Hepatitis C antibody positive.
4. Known HIV positivity (HIV testing will not be a requirement for this trial).
5. Serum creatinine > 500umol/l (consider MEPEX trial).
6. Immediately life-threatening organ manifestations (e.g. lung haemorrhage or dialysis dependence).
7. Previous malignancy (usually exclude unless agreed with trial co-ordinator).
8. Pregnancy or inadequate contraception if female.
9. Anti-GBM antibody positivity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 1998-02; Study Completion 2004-04

PRIMARY OUTCOMES:
Disease free period, time from remission to relapse or study end.

SECONDARY OUTCOMES:
Adverse events
Vasculitis Damage Index
Cumulative exposure to cyclophosphamide

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten de Groot, Study Chair — Klinikum Offenbach GmbH, Germany; Caroline OS Savage, Study Chair — University of Birmingham

REFERENCES:
- [Derived] Morgan MD, Szeto M, Walsh M, Jayne D, Westman K, Rasmussen N, Hiemstra TF, Flossmann O, Berden A, Hoglund P, Harper L; European Vasculitis Society. Negative anti-neutrophil cytoplasm antibody at switch to maintenance therapy is associated with a reduced risk of relapse. Arthritis Res Ther. 2017 Jun 7;19(1):129. doi: 10.1186/s13075-017-1321-1. PMID 28592297
- [Derived] de Groot K, Harper L, Jayne DR, Flores Suarez LF, Gregorini G, Gross WL, Luqmani R, Pusey CD, Rasmussen N, Sinico RA, Tesar V, Vanhille P, Westman K, Savage CO; EUVAS (European Vasculitis Study Group). Pulse versus daily oral cyclophosphamide for induction of remission in antineutrophil cytoplasmic antibody-associated vasculitis: a randomized trial. Ann Intern Med. 2009 May 19;150(10):670-80. doi: 10.7326/0003-4819-150-10-200905190-00004. PMID 19451574